CLINICAL TRIAL: NCT06510933
Title: Stability Effects After Heel Cups Orthopedics Treatment in Different BMI Index and Its Correlation to Physical Activity in Children. A Longitudinal Intervention Study
Brief Title: Stability Effects After Heel Cups Orthopedics Treatment in Different BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Vicenta Martínez Córcoles, Principal Investigator PhD, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCV/2017-2018/113
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Range of Motion
Keywords: BALANCE; HEEL CUPS; RANGE OF MOTION; PHYSICAL ACTIVITY
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Comparator: Heel Cup in muscle retraction (Experimental): The pattern will be performed 3 times per day (10 repetitions, 30 seconds each repetition). A daily Active Comparator: Heel Cup Group The heel cup will be 5mm high (Eva Shore 65) en 3 month and 6 month.
  Interventions: Device: Heel cups in different BMI index and its correlation to physical activity in children

INTERVENTIONS:
Device: Heel cups in different BMI index and its correlation to physical activity in children — Procedure: Group with muscle retraction will use a 5 millimeter heel cups in 3 and 6 months

SUMMARY:
Actual research relates Body mass Index (BMI) with postural changes in children and musculoskeletal disorders during growing period. BMI is widely used by clinicians and researchers due to easily capacity of application and scale classification patients in relation to their weight, the scale presents underweight, normal weight, overweight and obesity stages.

In paediatric context, underweight or overweight body mass in children negatively influences their posture, even in his adult life. Children with overweight and obesity shows less stability, and develop worse postural control, one of the demonstrated effects are the column alignment alteration and other bones structures. Elevated BMI are related to high differences in postural control, to elevated risk of pain, hypertension and musculoskeletal disorders. Underweight BMI is associated to less muscular mass and fat body composition, that are necessary to a correct posture, and contributes to increase probability of injuries.

The maintaining balance engages three systems, i.e., the vestibular system, vision, and proprioception. Some authors consider that postural stability develops between the ages 8 to 9. There are also papers arguing that the locomotor and postural model in 7-year-olds is similar to adults. Nevertheless, with new experiences and skills, it is possible to continue the development of all elements engaged in postural control, and keeping correct posture in children up to the age of 12 A good balance level and postural control is important in sport practice, to get high competition level efficiency in daily activities, and of course, in the clinic practice and rehabilitation.

Because of a stability loss off overweight in children, limited physical activity is established Posterior calf musculature and ankle has been shown to be involved in postural control in different studies. Likewise, the practice of physical activity induces changes in the infantile triceps suralis that generates improvements in postural control.

Currently, there are different paediatric pathologies for which heel cushions are prescribed as a treatment, such as Sever's disease leg, length discrepancy, relaxing and lenghtened calf muscles, but there is no evidence of stability effect of this treatment.

DETAILED DESCRIPTION:
A prospective intervention study was conducted in children before and after the application of heel cushions as a treatment for calf muscle retraction in various BMI conditions in children.

The design and progression of participants through the trial was conducted in accordance with the 22 CONSORT criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Children 8-12 years old
2. Regular sports practice
3. Decreased range of flexión

Exclusion Criteria:

1. Having neurological, vestibular, muscular, psychological or visual visual disease.
2. Traumatic pathology 12 months prior to the measurement (sprains, talalgias, etc.).
3. Diseases of balance or motor control.
4. Surgeries in the last 12 months.
5. Taking medications that may affect the neuromuscular system.
6. Sports practice in the last 48 hours.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Stabilometry | pre intervention, 3 months post intervention, 6 months post intervention
  The measurements were conducted in the primary school of participating schools at a temperature of 22 ◦C, in the same hour of the day. To assess participants' balance, the anthropometric position of the protocol proposed by the International Society for the Advancement of Cineatropometry (ISAK) was assigned: participants placed their mi Frankfort; the upper limbs remained relaxed throughout the body, with palms facing forward and thumbs separated from the rest of the toes, and were barefoot with feet externally rotated f 30 degrees and with a heel distance of 4cm. The children were wearing sports costumes to contribute their free movement. For stabilometry data collection will use an inertial measurement instrument called Gyko® It is a state-of-the-art device that allows to measure an objective assessment of acceleration, angular velocity and with an acquisition frequency of 100Hz
heel cups in muscle retraction | Pre intervention, 3 months post intervention, 6 months post intervention.
  Orthopaedic treatment of calf muscle retraction is defined as heel cup. A 5mm heel cup height was applied. Made of ethyl vinyl acetate material with a hard shore A 65º. The main function of a heel pad was to provide a slight change in heel elevation

SECONDARY OUTCOMES:
Lunge test | Pre intervention, 3 months post intervention, 6 months post intervention.
  To determine the dorsal flexion of the ankle, the Lunge Test was used. Through the Leg MOtion® system
Physical Activity Questionnaire for Children (PAQ-C) | Pre intervention, 3 months post intervention, 6 months post intervention
  The Spanish version of the Physical Activity Questionnaire for Children (PAQ-C) validated by Manchola- will be used to collect data on the type and amount of physical activity performed by the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Colegio Publico Cervantes, Munera, Albacete, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D Hondt E, Deforche B, De Bourdeaudhuij I, Lenoir M. Relationship between motor skill and body mass index in 5- to 10-year-old children. Adapt Phys Activ Q. 2009 Jan;26(1):21-37. doi: 10.1123/apaq.26.1.21. PMID 19246771
- [Result] D'Hondt E, Deforche B, De Bourdeaudhuij I, Gentier I, Tanghe A, Shultz S, Lenoir M. Postural balance under normal and altered sensory conditions in normal-weight and overweight children. Clin Biomech (Bristol). 2011 Jan;26(1):84-9. doi: 10.1016/j.clinbiomech.2010.08.007. Epub 2010 Sep 17. PMID 20850213
- [Result] Hermassi S, Ketelhut S, Konukman F, Ayari MA, Al-Marri S, Al Rawahi N, Bouhafs EG, Nigg CR, Schwesig R. Differences in Physical Activity, Sedentary Behavior, Health-Related Physical Performance Indices and Academic Achievement: A Comparative Study of Normal-Weight and Obese Children in Qatar. J Clin Med. 2024 Feb 13;13(4):1057. doi: 10.3390/jcm13041057. PMID 38398370
- [Result] Hommen JM, Batista JP, Bollheimer LC, Hildebrand F, Laurentius T, Siebers HL. Movement patterns during gait initiation in older adults with various stages of frailty: a biomechanical analysis. Eur Rev Aging Phys Act. 2024 Jan 13;21(1):1. doi: 10.1186/s11556-024-00335-w. PMID 38218828
- [Result] Barros WMA, da Silva KG, Silva RKP, Souza APDS, da Silva ABJ, Silva MRM, Fernandes MSS, de Souza SL, Souza VON. Effects of Overweight/Obesity on Motor Performance in Children: A Systematic Review. Front Endocrinol (Lausanne). 2022 Jan 20;12:759165. doi: 10.3389/fendo.2021.759165. eCollection 2021. PMID 35126307
- [Result] Pfeiffer M, Kotz R, Ledl T, Hauser G, Sluga M. Prevalence of flat foot in preschool-aged children. Pediatrics. 2006 Aug;118(2):634-9. doi: 10.1542/peds.2005-2126. PMID 16882817
- [Result] Nantel J, Mathieu ME, Prince F. Physical activity and obesity: biomechanical and physiological key concepts. J Obes. 2011;2011:650230. doi: 10.1155/2011/650230. Epub 2010 Nov 22. PMID 21113311
- [Result] Duncan MJ, Stanley M. Functional movement is negatively associated with weight status and positively associated with physical activity in british primary school children. J Obes. 2012;2012:697563. doi: 10.1155/2012/697563. Epub 2012 Mar 26. PMID 22545208
- [Result] Duncan MJ, Nevill A, Woodfield L, Al-Nakeeb Y. The relationship between pedometer-determined physical activity, body mass index and lean body mass index in children. Int J Pediatr Obes. 2010 Oct;5(5):445-50. doi: 10.3109/17477160903568421. PMID 20233151
- [Result] Mitchell UH, Johnson AW, Adamson B. Relationship between functional movement screen scores, core strength, posture, and body mass index in school children in Moldova. J Strength Cond Res. 2015 May;29(5):1172-9. doi: 10.1519/JSC.0000000000000722. PMID 25719919
- [Result] Martinez-Corcoles V, Nieto-Gil P, Ramos-Petersen L, Ferrer-Torregrosa J. Balance performance analysis after the COVID-19 quarantine in children aged between 8 and 12 years old: Longitudinal study. Gait Posture. 2022 May;94:203-209. doi: 10.1016/j.gaitpost.2022.03.019. Epub 2022 Mar 27. PMID 35366430